CLINICAL TRIAL: NCT06221267
Title: A Registry Study on Rimegepant for the Treatment of Migraine Participants in Guangdong-Hong Kong-Macao Greater Bay Area
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-1172-01
Record Dates: First submitted 2023-12-28; First posted 2024-01-24 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rimegepant — No intervention. The study will record the usage, timing, frequency, and dosage of rimegepant in a real-world clinical setting.

SUMMARY:
This study is a single-arm, prospective, multicenter, observational registry study. It plans to enroll 120 migraine patients who meet the inclusion criteria and are treated with rimegepant in selected hospital outpatient clinics in the Greater Bay Area. The main purpose of this study is to observe the effectiveness of rimegepant in treating migraines in a real-world clinical setting, including the impact of rimegepant on the quality of life, functioning, productivity status of migraine patients, and patients' satisfaction with the use of rimegepant in treating migraines.

ELIGIBILITY:
Inclusion Criteria:

* Participants with headaches that meet the diagnostic criteria for migraines according to the International Classification of Headache Disorders, 3rd edition (ICHD-3), with or without aura.
* Patients prescribed rimegepant by the attending physician for the treatment of migraines.
* Signed informed consent form.
* Age greater than 18 years.
* Not concurrently participating in other interventional clinical studies.

Exclusion Criteria:

* Patients diagnosed with secondary headaches.
* Patients with severe visual, auditory, language, intellectual, memory, consciousness impairments or other conditions that prevent them from completing the questionnaire and follow-up.
* Pregnant or lactating female patients.
* Patients deemed by the investigator as unsuitable for participation in the study or unable to complete the 4-week follow-up.
* Patients with a known history of hypersensitivity reactions to rimegepant or its components.
* Evidence in the medical history suggesting the presence of uncontrolled or unstable cardiovascular diseases (such as ischemic heart disease, coronary artery vasospasm, or cerebrovascular ischemia), or a history of myocardial infarction, acute coronary syndrome, percutaneous coronary intervention, cardiac surgery, stroke, or transient ischemic attack within the past 6 months before the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutively enroll 120 migraine patients who meet the inclusion criteria and are receiving treatment with rimegepant in selected outpatient clinics in the Guangdong-Hong Kong-Macao Greater Bay Area
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment Satisfaction Questionnaire for Medication (TSQM) | 4 weeks
  Treatment Satisfaction Questionnaire for Medication (TSQM) score for migraine patients' satisfaction with treatment of rimegepant
European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) | 4 weeks
  European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) score for the impact of rimegepant on the quality of life of migraine patients
Headache Impact Test-6 (HIT-6) | 4 weeks
  Headache Impact Test-6 (HIT-6) score for the impact of rimegepant on the functioning of migraine patients
Work Productivity and Activity Impairment-General Health (WPAI-GH) | 4 weeks
  Work Productivity and Activity Impairment-General Health (WPAI-GH) score for the impact of rimegepant on the productivity and work efficiency of migraine patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China